CLINICAL TRIAL: NCT00272415
Title: A Phase Ib, Open-Label, Multicenter Trial of Intravenous INO-1001 Plus Oral Temozolomide to Evaluate the Tolerability, Safety, and Pharmacokinetics in Subjects With Newly-Diagnosed or Recurrent Unresectable Stage III or Stage IV Melanoma
Brief Title: A Study of Intravenous INO-1001 Plus Oral Temozolomide to Evaluate Tolerability, Safety, and Pharmacokinetics in Patients With Melanoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Clinical Trials Posting Group, Genentech, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPC-06-2004; INO4136g
Record Dates: First submitted 2006-01-03; First posted 2006-01-06 (Estimated); Last update posted 2009-03-11 (Estimated); Status verified 2007-11

CONDITIONS: Melanoma
Keywords: INO4136g; inotek; Parp; Temodar
MeSH Terms: conditions — Melanoma; Deafness, Autosomal Recessive 53 | interventions — INO 1001; Temozolomide

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: INO-1001; Drug: temozolomide

INTERVENTIONS:
Drug: INO-1001 — Intravenous repeating dose
Drug: temozolomide — Oral repeating dose

SUMMARY:
This is a prospective, open-label, non-randomized, multicenter study in adults, aged eighteen (18) or older, with newly-diagnosed or recurrent unresectable Stage III or Stage IV melanoma. A maximum of 18 subjects will be enrolled in Stage 1 of this study. (Stage 1 completed enrollment in June 2006.) A maximum of 39 subjects will be enrolled in Stage 2 of this study.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven malignant melanoma with metastasis that is unresectable Stage III or Stage IV. Subjects with recurrent melanoma that is unresectable are also eligible
* Measurable indicator metastases
* Age 18 years or older
* ECOG status 0-2
* An interval at the time of enrollment of at least: a) 2 weeks since surgical resection (if conducted); b) 4 weeks since prior radiotherapy or chemotherapy, and c) 6 weeks since chemotherapy with a nitrosourea
* Hematocrit > 29%, ANC > 1500 cells/ul, platelets > 100,000 cells/ul
* Serum creatinine within the laboratory's upper limit of normal
* Serum AST and ALT ≤ 1.5 x the laboratory's upper limit of normal
* Subject signed informed consent prior to subject entry

Exclusion Criteria:

* Female patients who are pregnant or breast-feeding. Women of childbearing potential must have a negative serum or urine pregnancy test within 72 hours prior to administration of each cycle of the study drug regimen.
* Subjects of childbearing potential who are not willing or able to use an effective method of contraception, consisting of at least one-barrier method (e.g., condom and diaphragm), for the duration of the study and for at least 3 months after completing the treatment.
* Subjects previously treated with DTIC or TMZ
* Symptomatic central nervous metastases
* Concurrent severe and/or uncontrolled medical disease that could compromise participation in the study.
* Confirmed diagnosis of hepatitis or HIV infection
* Any medical, psychiatric, or social problem that might interfere with the performance, completion, and/or interpretation of the trial
* Patients who have had any surgery within two weeks prior to enrollment in this study, or who have not recovered from the side effects of this or any other therapy
* Patients unwilling to comply with the protocol or who in the judgment of the Principal Investigator are unable to abide by the rules of the protocol
* Subjects who have received a potent CYP3A4 inhibitor or inducer orally or parenterally within approximately 14 days prior to enrollment
* Subjects who have received amiodarone within 30 days of study drug administration
* History of hypersensitivity reaction to more than three (3) drugs or to mannitol
* Patients who have received any investigational study agent within 30 days of Day 1 of Cycle 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2005-10

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) or recommended Phase II dose of INO-1001 to be used in combination with TMZ | Length of study
Pharmacokinetic (PK) profile of intravenous INO-1001 | Length of study
Safety and tolerability of combined therapy with oral temozolomide (TMZ) and intravenous INO-1001 | Length of study

SECONDARY OUTCOMES:
Safety of repeat dosing | Length of study
Pharmacodynamic (PD) activity of intravenous INO-1001 | Length of study
Response | Length of study
Progression-free survival | Length of study
Overall survival | Length of study

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Low, M.D., Ph.D., Study Director — Genentech, Inc.